CLINICAL TRIAL: NCT00967161
Title: 3D Motion Analysis of Evolution Medial Pivot Knee VS Posterior Stabilized Knee Arthroplasty for Osteoarthritis of the Knee.Feasibility Pilot for a Prospective Randomized Controlled Trial.
Brief Title: Motion Analysis of EMP Knee Versus Posterior Stabilized Knee Arthroplasty for Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: OHREB 2009-240-01H
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Arthropathy of Knee Joint
Keywords: knee replacement motion analysis
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evolution Medial Pivot Knee (Experimental): 20 Patients will receive the EMP Knee Implant
  Interventions: Procedure: Total Knee Arthroplasty; Procedure: Motion analysis
- Triathlon PS Knee (Active Comparator): 20 Patients will receive the Triathlon PS Knee
  Interventions: Procedure: Total Knee Arthroplasty; Procedure: Motion analysis

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Total Knee Arthroplasty
  Other Names: non applicable
Procedure: Motion analysis — Motion analysis (Gait/EMG during walking and functional tasks)
  Other Names: non applicable

SUMMARY:
The purpose of the current study is to analyze and compare the lower-limb joint motions and muscle activation patterns during activities of daily living as well as self reported health related functional outcomes for patients with osteoarthritis of the knee undergoing one of two types of knee replacements: the Evolution Medial Pivot knee (Wright Medical) or the Triathlon Posterior Stabilized (PS) knee (Stryker Orthopaedics).

DETAILED DESCRIPTION:
Inclusion:

40 patients between the ages of 50 and 75 yrs undergoing unilateral total knee replacement for non-inflammatory degenerative osteoarthritis will participate, as well as 10 control participants will be recruited from the general population for the present study matching to experimental groups for age, gender and BMI.

Patients who do not meet any exclusion criteria.

Exclusion:

Potential participants for the control group will be asked if they have had degenerative osteoarthritis of lower-limb joints (hip, knee and ankle) and if they have they will be excluded.

Exclusion for patient group

1. Patients suffering from any other lower-limb joint disorders other than the one for which total knee arthroplasty.
2. Patients with any other joint replacement in the ipsilateral and contralateral limb.
3. Patients with evidence of active infection.
4. Patients with neurologic or musculoskeletal disease that may adversely affect gait, weight-bearing or quadriceps function.
5. Patients with neuropathic joints.
6. Patients requiring structural bone grafts.
7. Patients with a documented allergy to cobalt chromium molybdenum.
8. Patient with a BMI larger than 30 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* 40 patients between the ages of 50 and 75 yrs undergoing unilateral total knee replacement for non-inflammatory degenerative osteoarthritis will participate, as well as 10 control participants will be recruited from the general population for the present study matching to experimental groups for age, gender and BMI.Patients who do not meet any exclusion criteria.

Exclusion Criteria:

* Potential participants for the control group will be asked if they have had degenerative osteoarthritis of lower-limb joints (hip, knee and ankle) and if they have they will be excluded.

Exclusion for patient group

1. Patients suffering from any other lower-limb joint disorders other than the one for which total knee arthroplasty.
2. Patients with any other joint replacement in the ipsilateral and contralateral limb.
3. Patients with evidence of active infection.
4. Patients with neurologic or musculoskeletal disease that may adversely affect gait, weight-bearing or quadriceps function.
5. Patients with neuropathic joints.
6. Patients requiring structural bone grafts.
7. Patients with a documented allergy to cobalt chromium molybdenum.
8. Patient with a BMI larger than 30 kg/m2.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The motion analysis assessments of the knee | pre-op,6,12 months following surgery

SECONDARY OUTCOMES:
Questionnaires: RAND-36, Knee injury and Osteoarthritis Outcome Score (KOOS) and Satisfaction survey. | pre-op,6,12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Dervin, MD,MSc,FRCSC, Principal Investigator — OHRI / The Ottawa Hospital/ University of Ottawa
Locations (1):
- The Ottawa General Hospital, Ottawa, Ontario, Canada